CLINICAL TRIAL: NCT03508700
Title: A 40-week Open-Label Extension Study to Evaluate TNX-102 SL 5.6 mg Taken Daily at Bedtime in Patients With PTSD
Brief Title: A 40-week Study to Evaluate TNX-102 SL 5.6 mg Taken Daily at Bedtime in Patients With PTSD
Acronym: P306
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-P306
Record Dates: First submitted 2018-04-12; First posted 2018-04-26 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: PTSD
Keywords: TNX-102 SL; Bedtime; Sublingual; Safety; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TNX-102 SL 5.6 mg (Experimental): 2 tablets of TNX-102 SL 2.8 mg taken simultaneously and sublingually (under the tongue) each day at bedtime starting on Day 0 for 40 weeks
  Interventions: Drug: TNX-102 SL 5.6 mg

INTERVENTIONS:
Drug: TNX-102 SL 5.6 mg — cyclobenzaprine HCl sublingual tablets

SUMMARY:
Evaluate the long-term safety of TNX-102 SL 5.6 mg taken daily at bedtime over an additional 40 weeks in patients with PTSD who have participated in a double-blind lead-in study and completed an initial 12-week open-label extension study (TNX-CY-P303).

DETAILED DESCRIPTION:
This is an open-label, extension trial designed to evaluate safety over 40 additional weeks of TNX-102 SL therapy taken daily at bedtime for the treatment of PTSD.

The study will consist of 5 in-clinic study visits, including Baseline Visit 1 (Day 0, which is anticipated to be the same visit as the last visit of the 12-week open-label extension study TNX-CY-P303), followed by in-clinic visits after 7, 16, 28 and 40 weeks of open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed a double-blind lead-in HONOR study and a 12-week open-label extension study P303 and is judged by the investigator as reasonably compliant, with at least 60% compliance with study medication usage (based on drug accountability).
* The patient has provided written informed consent to participate in this extension study.
* The patient met all prior inclusion and exclusion requirements for the double-blind lead-in HONOR study, or the site received medical monitor approval for the patient to remain in the lead-in study after the retrospective discovery of an entry violation that did not pose any threat to the patient's safety or well-being.
* During the course of the lead-in HONOR study or 12-week open-label extension P303 study, the patient has had no intervening medical conditions including pregnancy, clinically significant increase in suicidal ideation (plan or intent) or significant worsening of depression, newly arising clinically significant abnormal laboratory tests, or any clinically significant, uncontrolled, or unstable medical or surgical condition that could affect the patient's ability to participate in the study or potentially compromise the patient's well-being during the study.
* The patient does not require treatment with a potent (strong) cytochrome P450 subtype 3A4 (CYP3A4) inhibitor, or St. John's wort.
* The patient is willing to refrain from use of all other formulations of cyclobenzaprine for the duration of the study.
* The patient is willing to refrain from use of monoamine oxidase inhibitors for the duration of the study.
* Female patients of childbearing potential continue to agree to practice one of the medically acceptable methods of birth control detailed in the lead-in study.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Little Rock, Little Rock, Arkansas
  - Beverly Hills, Beverly Hills, California
  - Oceanside, Oceanside, California
  - Orange, Orange, California
  - Temecula, Temecula, California
  - Colorado Springs, Colorado Springs, Colorado
  - Norwich, Norwich, Connecticut
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - New Bedford, New Bedford, Massachusetts
  - Las Vegas, Las Vegas, Nevada
  - Cedarhurst, Cedarhurst, New York
  - New York, New York, New York
  - Canton, Canton, Ohio
  - Cincinnati, Cincinnati, Ohio
  - Oklahoma City, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - TNX-102 SL: This group received placebo in the lead-in double blind study TNX-CY-P301, and received TNX-102-SL 5.6 mg in this open label study TNX-CY-P306.
- TNX-102 SL - TNX-102 SL: This group received TNX-102 SL 5.6 mg in the lead-in double blind study TNX-CY-P301, and received TNX-102 SL 5.6mg in this open label study TNX-CY-P306.
Period: Overall Study
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
Started | 49 | 44
Completed | 28 | 29
Not Completed | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL | Total
Number analyzed (Participants) | 49 | 44 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (9.29) | 34.5 (7.91) | 36.8 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 41 | 41 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 41 | 41 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 9 | 9 | 18
  White | 31 | 26 | 57
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 49 | 44 | 93

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Newly Emergent Adverse Events
Description: Evaluate the incidence of newly emergent adverse events over an additional 40 weeks of treatment with TNX-102 SL 5.6 mg in patients with PTSD who have participated in a double-blinded lead-in study. Adverse events will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized overall and by preferred term and system organ class. Serious AEs and AEs leading to discontinuation of study drug will also be summarized.
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
Number analyzed (Participants) | 49 | 44
Participants | 26 | 19

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/44
Other Adverse Events (participants affected / at risk) | 6/49 | 2/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - TNX-102 SL (N=49) | TNX-102 SL - TNX-102 SL (N=44)
Hypoaesthesia oral (Gastrointestinal disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03508700/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03508700/SAP_001.pdf